CLINICAL TRIAL: NCT02307760
Title: Evaluation of Two Human Milk Fortifiers in Preterm Infants
Brief Title: Evaluation of Human Milk Fortifiers in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AL16
Record Dates: First submitted 2014-12-01; First posted 2014-12-04 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Infant Growth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Human Milk Fortifier A (Active Comparator): Acidified processing method.
  Interventions: Other: Human Milk Fortifier A
- Study Human Milk Fortifier B (Experimental): Non-acidified processing method.
  Interventions: Other: Human Milk Fortifier B

INTERVENTIONS:
Other: Human Milk Fortifier A — Acidified concentrated liquid human milk fortifier
  Arms: Study Human Milk Fortifier A
Other: Human Milk Fortifier B — Non-acidified concentrated liquid human milk fortifier
  Arms: Study Human Milk Fortifier B

SUMMARY:
The purpose of this study is to assess growth of preterm infants fed human milk supplemented with one of two commercially available human milk fortifiers.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight of 700 g-1500 g.
* ≤ 32 weeks and 0 days GA at birth.
* Appropriate for GA (AGA).
* Enteral feeding of human milk initiated by 21 days of life (birth date is day of life 0).
* Mother agrees to provide human milk as the exclusive feeding during the study period; use of donor milk is permitted if the plan is that it will be fortified.
* Parent(s) agrees to allow infant to receive both human milk and HMF.
* Singleton or twin births only.

Exclusion Criteria:

* Enteral feeding of preterm infant formula or HMF for > 7 days.
* Expected to be transferred to another facility and will not be able to be followed for at least 15 days.
* Serious congenital abnormalities or underlying disease that may affect growth and development.
* 5 minute APGAR ≤ 4.
* Steroids used at the time of randomization.
* Grade III or IV periventricular/intraventricular hemorrhage (PVH/IVH).
* Mechanical ventilator dependence.
* Maternal incapacity: including maternal cocaine or alcohol abuse during pregnancy or current, or if the mother or infant is currently receiving treatment consistent with HIV therapy.
* Infant has a history of major surgery (intra-thoracic or intra-abdominal procedures or other surgery requiring general anesthesia).
* Asphyxia defined as progressive hypoxemia and hypercapnia with significant metabolic acidemia characterized by APGAR score <3 at 10 minutes, seizures within the first 12 hours of life, or a cord blood gas < 7.0 and seizures and/or severe tonic abnormalities in the first 12 hours of life (24).
* Confirmed necrotizing enterocolitis (Bell's Stage II or III, Appendix J) or confirmed sepsis (positive culture requiring antibiotic treatment).
* Infant has any other condition that, in the opinion of the investigator, precludes participation in the study.
* Participation in another study that has not been approved as a concomitant study by AN.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Weight Gain | Study Day 1 to Study Day 29 (or discharge, whichever happens first)
  scale measurement g/kg/d

SECONDARY OUTCOMES:
Gastrointestinal Tolerance | Study Day 1 to Study Day 29 (or discharge, whichever happens first)
  healthcare professional completed questionnaire
Length | Study Day 1 to Study Day 29 (or discharge, whichever happens first)
  measured cm/wk
Head Circumference | Study Day 1 to Study Day 29 (or discharge, whichever happens first)
  measured cm/wk

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Barrett-Reis, PhD, RD, Study Chair — Abbott Nutrition
Locations (18):
- United States (18):
  - University of South Alabama Children's and Women's Hospital, Mobile, Alabama
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Yale University, New Haven, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - South Miami Hospital, Miami, Florida
  - All Children's Hospital / Johns Hopkins, St. Petersburg, Florida
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Louisville, Louisville, Kentucky
  - Cohen Children's Medical Center of NY at North Shore, Manhasset, New York
  - Cohen Children's Medical Center of NY, New Hyde Park, New York
  - Duke University Medical Center, Durham, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Doctors Hospital at Renaissance/Women's Hospital at Renaissance, Edinburg, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Health and Education Institute, Fort Worth, Texas
  - North Central Baptist Hospital, San Antonio, Texas
  - Wheaton Franciscan Heathcare Inc.- St. Joseph, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paul M, Partridge J, Barrett-Reis B, Ahmad KA, Machiraju P, Jayapalan H, Schanler RJ. Metabolic Acidosis in Preterm Infants is Associated with a Longer Length of Stay in the Neonatal Intensive Care Unit. Pharmacoecon Open. 2020 Sep;4(3):541-547. doi: 10.1007/s41669-020-00194-y. PMID 31975350
- [Derived] Schanler RJ, Groh-Wargo SL, Barrett-Reis B, White RD, Ahmad KA, Oliver J, Baggs G, Williams L, Adamkin D. Improved Outcomes in Preterm Infants Fed a Nonacidified Liquid Human Milk Fortifier: A Prospective Randomized Clinical Trial. J Pediatr. 2018 Nov;202:31-37.e2. doi: 10.1016/j.jpeds.2018.07.005. Epub 2018 Sep 5. PMID 30195561